CLINICAL TRIAL: NCT01764906
Title: The Clinical Study to Evaluate the Efficacy and Safety of Novosis in Posterolateral Fusion
Brief Title: The Clinical Study of Novosis in Posterolateral Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: BioAlpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA06-CP01
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2013-01

CONDITIONS: Posterolateral Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novosis (Experimental): Bongros/rhBMP-2
  Interventions: Device: Novosis
- Iliac crest bone graft (Active Comparator): Iliac crest bone graft
  Interventions: Procedure: Iliac crest bone graft

INTERVENTIONS:
Device: Novosis
  Arms: Novosis
Procedure: Iliac crest bone graft
  Arms: Iliac crest bone graft

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Novosis in posterolateral fusion

ELIGIBILITY:
Inclusion Criteria:

* 18~80 aged patients needed single-level posterolateral fusion at L1~S1
* A subject who provided written informed consent to participate in this study

Exclusion Criteria:

* Patients with BMD T-score < -3.0
* Women who are pregnant or plan to be pregnant within study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Fusion grade by CT assessments after surgery | 24 weeks

SECONDARY OUTCOMES:
Fusion grade by Radiographic assessments after surgery | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea